CLINICAL TRIAL: NCT02735057
Title: Phase I-II Study Chemoradiation in Elderly Patients With Oesophagus Cancer
Brief Title: Chemoradiotherapy in Elderly Patients With Oesophagus Cancer
Acronym: OSAGE
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N/2014/68
Record Dates: First submitted 2016-03-18; First posted 2016-04-12 (Estimated); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Oesophagus Cancer; Elderly Patients
Keywords: oesophagus cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Phase I (Experimental): * for chemotherapy 3 levels: 50%, 75% and 100% of the standard Dutch dose (carboplatin AUC 2 and paclitaxel 50 mg/m2)
  * for radiotherapy 3 levels: 41.4 Gy/1.8 Gy/f; 45 Gy/1.8 Gy/f; 50.4 Gy/1.8 Gy/f basel level being : 41.4 Gy and 50% of standard CT doses The phase I is conducted with increasing doses of each component with 9 levels.
  Interventions: Drug: Carboplatin

INTERVENTIONS:
Drug: Carboplatin
  Other Names: Paclitaxel

SUMMARY:
Management of elderly patient with cancer is a therapeutic challenge and a public health problem. The mean age of esophageal cancer is 64.5 years and 72.1 years in men and women respectively. Surgery is a standard treatment reserved to about 30 % of patients. The other 70 % are considered unfit for surgery for various reasons, including ageing.

Chemoradiotherapy (CRT) is standard treatment for patients with esophageal cancer unfit for surgery. The validated treatment scheme is external beam radiotherapy (EBRT) 50 Gy over 5 weeks combined with cisplatin and 5FU infusion. However it induces high rates of severe and life threatening toxicities: grade 3 haematologic and esophageal mucositis of 20 and 25 % respectively, in patients with a median age of 64 years. CRT has not been properly evaluated in patients more than 75 years, and other combined chemotherapy are challenging.

DETAILED DESCRIPTION:
Choice of the combined chemotherapy Carboplatin and taxanes delivered concurrently to radiotherapy is attractive. A Dutch randomized study (Cross trial) compared preoperative CRT to surgery in 368 patients with T1-T3 and N0N1. In the preoperative CRT group, patients received 41.4 Gy by EBRT over 5 weeks combined with carboplatin (AUC 2) and paclitaxel (50 mg/m2). A 30 % tumor sterilization rate and a reduction of metastasis considered a distant effect of chemotherapy were observed. The 5-year survival was statistically better with CRT group. The preoperative CRT was well tolerated and few acute toxicities were observed. Intriguingly, in a French randomized study, conducted in less locally advanced disease, the combination of 45 Gy and 5 FU infusion and Cisplatin did not induce more tumor sterilization rate, suggesting carboplatine/paclitaxel is more effective than 5FU/cisplatin in CRT.

Study design Since the optimal doses of each component radiotherapy- carboplatin - paclitaxel are unknown, we plan to conduct a phase I/II study

* Phase I: the objective is to determine the maximum tolerated dose (MTD) and recommended doses for phase II (RP2D) of each component considering the treatment scheme of Dutch study as reference:

  * for chemotherapy 3 levels: 50%, 75% and 100% of the standard Dutch dose (carboplatin AUC 2 and paclitaxel 50 mg/m2)
  * for radiotherapy 3 levels: 41.4 Gy/1.8 Gy/f; 45 Gy/1.8 Gy/f; 50.4 Gy/1.8 Gy/f basel level being : 41.4 Gy and 50% of standard CT doses The phase I is conducted with increasing doses of each component with 9 levels.
* Phase II: after the determination of RP2D of each component, the study is continued as a phase II in order to assess tumor response Secondary objectives: Quality of life, progression free and overall survivals

ELIGIBILITY:
Inclusion Criteria:

* Esophageal cancer, squamous and adenocarcinoma types, T1-3, N0-1, M1a (TNM 6th),
* age > 75 years,
* WHO status < 2, Balducci 1, adequate bone marrow reserve, normal renal and hepatic function.

Exclusion Criteria:

* age < 75 years

Ages: 75 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2016-04-04 (Actual); Primary Completion 2028-11-16 (Estimated); Study Completion 2029-05-16 (Estimated)

PRIMARY OUTCOMES:
maximum tolerated dose (MTD) | 1 months after the end of the treatment
  the objective is to determine the maximum tolerated dose (MTD) and recommended doses for phase II.The phase I is conducted with increasing doses of each component with 9 levels.Step definitively stopped in case of any grade ≥ 3 or severe acute toxicities. In case a step is definitively stopped, add 3 more patients to the precedent step.
  Quality assurance

SECONDARY OUTCOMES:
Quality of life | 3 years
  EORTC QLQ-C30,
Quality of life | 3 years
  ELD14
progression free survival | 3 years
overall survival | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire de Besançon, Besançon, France

REFERENCES:
- [Derived] Servagi-Vernat S, Crehange G, Bonnetain F, Mertens C, Brain E, Bosset JF. Chemoradiation in elderly esophageal cancer patients: rationale and design of a phase I/II multicenter study (OSAGE). BMC Cancer. 2017 Jul 13;17(1):483. doi: 10.1186/s12885-017-3465-4. PMID 28705182